CLINICAL TRIAL: NCT00542178
Title: Action to Control Cardiovascular Risk in Diabetes (ACCORD) Eye Study
Brief Title: Evaluating How the Treatments in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Study Affect Diabetic Retinopathy (The ACCORD Eye Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 509; N01 HC095178-19; N01HC095178 (NIH)
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2016-10

CONDITIONS: Diabetic Retinopathy
Keywords: Type 2 Diabetes Mellitus; Cardiovascular Diseases
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Hypoglycemic Agents; Fenofibrate; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Intensive glycemia control (Experimental): A strategy of intensive glycemia treatment to HbA1c less than 6%
  Interventions: Drug: Hypoglycemic Agents
- Standard glycemia control (Active Comparator): A strategy of multiple drugs to treat HbA1c to 7.0% - 7.9%
  Interventions: Drug: Standard glycemia control
- Intensive BP control (Experimental): A strategy of BP treatment for SBP less than 120 mm Hg
  Interventions: Drug: Intensive BP treatment
- Standard BP control (Active Comparator): A strategy of BP treatment for SBP less than 140 mm Hg
  Interventions: Drug: Standard BP control
- Fibrate (Experimental): Blinded fenofibrate + simvastatin 20-40 mg/d
  Interventions: Drug: Fenofibrate; Drug: Simvastatin
- Fibrate Placebo (Placebo Comparator): Blinded placebo + simvastatin 20-40 mg/d
  Interventions: Drug: Simvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Hypoglycemic Agents — Multiple drugs including insulins and oral hypoglycemia agents for HbA1c less than 6%
  Arms: Intensive glycemia control
Drug: Standard glycemia control — A strategy of glycemia drugs for HbA1c 7% - 7.9%
  Arms: Standard glycemia control
Drug: Intensive BP treatment — A strategy of multiple BP agents to reduce SBP less than 120 mm Hg
  Arms: Intensive BP control
Drug: Standard BP control — A strategy of BP drugs for SBP less than 140 mm Hg
  Arms: Standard BP control
Drug: Fenofibrate — Blinded fenofibrate
  Arms: Fibrate
Drug: Simvastatin — Simvastatin 20-40 mg/d
  Arms: Fibrate; Fibrate Placebo
Drug: Placebo — Placebo
  Arms: Fibrate Placebo

SUMMARY:
Diabetic retinopathy (DR) is an eye disease that can occur in people with diabetes and can cause poor vision or blindness. The Action to Control Cardiovascular Risk in Diabetes (ACCORD) study is examining the effect of various treatments on cardiovascular disease in people with diabetes. This current study will examine the effects of the ACCORD treatments on the progression of DR in people participating in the ACCORD study.

DETAILED DESCRIPTION:
DR is the most common diabetic eye disease and is the leading cause of blindness in adults in the United States. It is caused by damage to the blood vessels of the retina, which is the light-sensitive outer layer of the eye. Retinal blood vessels are often affected by the high blood sugar levels associated with diabetes. Older people have an increased risk of developing DR; however, DR is likely to occur earlier and be more severe in anyone who has poorly controlled diabetes. Almost everyone who has had diabetes for more than 30 years will eventually show signs of DR. Symptoms of DR include poor night vision, seeing spots in front of the eyes, blurred vision, and blindness. The ACCORD study is a study that is examining the effects of different treatments on cardiovascular disease in people with diabetes. Participants in the ACCORD study will receive one of eight different combinations of treatment, including blood sugar control, blood pressure control, and cholesterol-controlling medication. This study will enroll participants in the ACCORD study and will examine the effects of the study treatments on DR. The results from this study may be used to develop new treatments to help prevent diabetes-related blindness.

Study visits will occur at baseline and Year 4. At each study visit, participants will have an eye exam and specialized fundus photographs taken of the back of the eye and retina.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the ACCORD study

Exclusion Criteria:

* Has had laser photocoagulation for DR
* Has had vitrectomy surgery for DR

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3472 (Actual)
Dates: Start 2003-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter T. Ambrosius, PhD, Principal Investigator — Wake Forest University Health Sciences; Emily Y. Chew, MD, Principal Investigator — National Eye Institute (NEI)
Locations (7):
- United States (6):
  - The Berman Center for Clinical Research, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Veterans Affairs, Memphis, Tennessee
  - University of Washington, Seattle, Washington
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Chew EY, Ambrosius WT, Howard LT, Greven CM, Johnson S, Danis RP, Davis MD, Genuth S, Domanski M; ACCORD Study Group. Rationale, design, and methods of the Action to Control Cardiovascular Risk in Diabetes Eye Study (ACCORD-EYE). Am J Cardiol. 2007 Jun 18;99(12A):103i-111i. doi: 10.1016/j.amjcard.2007.03.028. Epub 2007 Apr 13. PMID 17599420
- [Result] ACCORD Study Group; ACCORD Eye Study Group; Chew EY, Ambrosius WT, Davis MD, Danis RP, Gangaputra S, Greven CM, Hubbard L, Esser BA, Lovato JF, Perdue LH, Goff DC Jr, Cushman WC, Ginsberg HN, Elam MB, Genuth S, Gerstein HC, Schubart U, Fine LJ. Effects of medical therapies on retinopathy progression in type 2 diabetes. N Engl J Med. 2010 Jul 15;363(3):233-44. doi: 10.1056/NEJMoa1001288. Epub 2010 Jun 29. PMID 20587587
- [Derived] Do DV, Han G, Abariga SA, Sleilati G, Vedula SS, Hawkins BS. Blood pressure control for diabetic retinopathy. Cochrane Database Syst Rev. 2023 Mar 28;3(3):CD006127. doi: 10.1002/14651858.CD006127.pub3. PMID 36975019
- [Derived] Action to Control Cardiovascular Risk in Diabetes Follow-On (ACCORDION) Eye Study Group and the Action to Control Cardiovascular Risk in Diabetes Follow-On (ACCORDION) Study Group. Persistent Effects of Intensive Glycemic Control on Retinopathy in Type 2 Diabetes in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Follow-On Study. Diabetes Care. 2016 Jul;39(7):1089-100. doi: 10.2337/dc16-0024. Epub 2016 Jun 11. PMID 27289122
- [Derived] Chew EY, Davis MD, Danis RP, Lovato JF, Perdue LH, Greven C, Genuth S, Goff DC, Leiter LA, Ismail-Beigi F, Ambrosius WT; Action to Control Cardiovascular Risk in Diabetes Eye Study Research Group. The effects of medical management on the progression of diabetic retinopathy in persons with type 2 diabetes: the Action to Control Cardiovascular Risk in Diabetes (ACCORD) Eye Study. Ophthalmology. 2014 Dec;121(12):2443-51. doi: 10.1016/j.ophtha.2014.07.019. Epub 2014 Aug 29. PMID 25172198
- [Derived] Wong TY, Simo R, Mitchell P. Fenofibrate - a potential systemic treatment for diabetic retinopathy? Am J Ophthalmol. 2012 Jul;154(1):6-12. doi: 10.1016/j.ajo.2012.03.013. PMID 22709833
- [Derived] Ambrosius WT, Danis RP, Goff DC Jr, Greven CM, Gerstein HC, Cohen RM, Riddle MC, Miller ME, Buse JB, Bonds DE, Peterson KA, Rosenberg YD, Perdue LH, Esser BA, Seaquist LA, Felicetta JV, Chew EY; ACCORD Study Group. Lack of association between thiazolidinediones and macular edema in type 2 diabetes: the ACCORD eye substudy. Arch Ophthalmol. 2010 Mar;128(3):312-8. doi: 10.1001/archophthalmol.2009.310. PMID 20212201
- See also: Click here for the ACCORD Study Web site — http://www.accordtrial.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the ACCORD Eye study was restricted to participants recruited as part of the Action to Control Cardiovascular Risk in Diabetes (ACCORD) study. The ACCORD Eye study began in October 2003, with 3472 participants enrolled by February 2006.
Pre-assignment Details: All participants were enrolled in either the intensive or standard glycemia control arms. In addition to inclusion in the glycemia control part of the trial, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo).
Groups:
- Intensive Glycemia Control & Intensive Blood Pressure Control: Intensive Glycemia Control: A strategy of intensive glycemia treatment to HbA1c less than 6%
  Intensive Blood Pressure Control: A strategy of BP treatment for SBP less than 120 mm Hg
- Standard Glycemia Control & Intensive Blood Pressure Control: Standard Glycemia Control: A strategy of multiple drugs to treat HbA1c to 7.0% - 7.9%
  Intensive Blood Pressure Control: A strategy of BP treatment for SBP less than 120 mm Hg
- Intensive Glycemia Control & Standard Blood Pressure Control: Intensive Glycemia Control: A strategy of intensive glycemia treatment to HbA1c less than 6%
  Standard Blood Pressure Control: A strategy of BP treatment for SBP less than 140 mm Hg
- Standard Glycemia Control & Standard Blood Pressure Control: Standard Glycemia Control: A strategy of multiple drugs to treat HbA1c to 7.0% - 7.9%
  Standard Blood Pressure Control: A strategy of BP treatment for SBP less than 140 mm Hg
- Intensive Glycemia Control & Fibrate: Intensive Glycemia Control: A strategy of intensive glycemia treatment to HbA1c less than 6%
  Fibrate: Blinded fenofibrate + simvastatin 20-40 mg/d
- Standard Glycemia Control & Fibrate: Standard Glycemia Control: A strategy of multiple drugs to treat HbA1c to 7.0% - 7.9%
  Fibrate: Blinded fenofibrate + simvastatin 20-40 mg/d
- Intensive Glycemia Control & Fibrate Placebo: Intensive Glycemia Control: A strategy of intensive glycemia treatment to HbA1c less than 6%
  Fibrate Placebo: Blinded placebo + simvastatin 20-40 mg/d
- Standard Glycemia Control & Fibrate Placebo: Standard Glycemia Control: A strategy of multiple drugs to treat HbA1c to 7.0% - 7.9%
  Fibrate Placebo: Blinded placebo + simvastatin 20-40 mg/d
Period: Overall Study
Arm/Group | Intensive Glycemia Control & Intensive Blood Pressure Control | Standard Glycemia Control & Intensive Blood Pressure Control | Intensive Glycemia Control & Standard Blood Pressure Control | Standard Glycemia Control & Standard Blood Pressure Control | Intensive Glycemia Control & Fibrate | Standard Glycemia Control & Fibrate | Intensive Glycemia Control & Fibrate Placebo | Standard Glycemia Control & Fibrate Placebo
Started | 390 | 412 | 382 | 370 | 464 | 495 | 493 | 466
Completed | 315 | 332 | 308 | 308 | 400 | 406 | 406 | 381
Not Completed | 75 | 80 | 74 | 62 | 64 | 89 | 87 | 85
Not completed — did not complete year 4 follow-up | 75 | 80 | 74 | 62 | 64 | 89 | 87 | 85

BASELINE CHARACTERISTICS:
Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Glycemia Control | Standard Glycemia Control | Intensive BP Control | Standard BP Control | Fibrate | Fibrate Placebo | Total
Number analyzed (Participants) | 1429 | 1427 | 647 | 616 | 806 | 787 | 5712
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (6.4) | 61.5 (6.3) | 61.3 (6.1) | 61.5 (6.6) | 61.9 (6.2) | 61.5 (6.5) | 61.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  Participants
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study: Female | 538 | 552 |  |  |  |  | 1090
    Glycemic Control Study: Male | 891 | 875 |  |  |  |  | 1766
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies: Female |  |  | 310 | 279 | 247 | 254 | 1090
    Blood Pressure and Lipid Studies: Male |  |  | 337 | 337 | 559 | 533 | 1766
Duration of diabetes [Mean (Standard Deviation); unit: year] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  year
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 9.8 (7.1) | 10.1 (7.2) |  |  |  |  | 10.0 (7.1)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 10.1 (7.0) | 10.3 (7.5) | 9.7 (6.8) | 9.8 (7.2) | 10.0 (7.1)
Previous cardiovascular event [Count of Participants; unit: Participants] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  Participants
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study: Previous cardiovascular event | 452 | 443 |  |  |  |  | 895
    Glycemic Control Study: No previous cardiovascular event | 977 | 984 |  |  |  |  | 1961
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies: Previous cardiovascular event |  |  | 180 | 197 | 263 | 255 | 895
    Blood Pressure and Lipid Studies: No previous cardiovascular event |  |  | 467 | 419 | 543 | 532 | 1961
Race [Count of Participants; unit: Participants] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  Participants
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study: Nonwhite race | 427 | 433 |  |  |  |  | 860
    Glycemic Control Study: White race | 1002 | 994 |  |  |  |  | 1996
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies: Nonwhite race |  |  | 203 | 201 | 222 | 234 | 860
    Blood Pressure and Lipid Studies: White race |  |  | 444 | 415 | 584 | 553 | 1996
Glycated hemoglobin [Mean (Standard Deviation); unit: percent] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  percent
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 8.2 (1.0) | 8.3 (1.0) |  |  |  |  | 8.2 (1.0)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 8.4 (1.1) | 8.2 (1.0) | 8.2 (1.0) | 8.2 (1.0) | 8.2 (1.0)
Cholesterol (HDL) [Mean (Standard Deviation); unit: mg/dl] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  mg/dl
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 42.0 (11.4) | 41.9 (11.1) |  |  |  |  | 41.9 (11.3)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 46.3 (12.8) | 46.31 (13.8) | 38.6 (7.8) | 38.5 (7.9) | 41.9 (11.3)
Cholesterol (LDL) [Mean (Standard Deviation); unit: mg/dl] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  mg/dl
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 100.8 (33.4) | 100.7 (32.1) |  |  |  |  | 100.7 (32.7)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 107.4 (37.0) | 104.1 (33.5) | 96.5 (29.7) | 97.0 (30.1) | 100.7 (32.7)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  mg/dl
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 196.1 (157.8) | 194 (167.3) |  |  |  |  | 195.1 (162.6)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 200.7 (175.5) | 204.7 (240.3) | 190.1 (111.3) | 187.9 (112.4) | 195.1 (162.6)
Systolic Blood pressure [Mean (Standard Deviation); unit: mm Hg] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  mm Hg
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 134.3 (16.6) | 134.7 (17.4) |  |  |  |  | 134.5 (17.0)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 138.0 (16.7) | 139.0 (14.7) | 131.5 (17.0) | 131.1 (17.5) | 134.5 (17.0)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  mm Hg
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 74.9 (10.3) | 75.0 (10.6) |  |  |  |  | 74.9 (10.5)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 76.3 (10.5) | 76.8 (9.9) | 73.7 (10.5) | 73.6 (10.5) | 74.9 (10.5)
Urinary albumin:creatinine ratio [Mean (Standard Deviation); unit: albumin (mg/dL): creatinin (g/dL)] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  albumin (mg/dL): creatinin (g/dL)
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 69.5 (2228.9) | 74.0 (275.3) |  |  |  |  | 71.8 (253.1)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 62.5 (197.6) | 79.2 (269.9) | 62.3 (180.2) | 83.2 (331.5) | 71.8 (253.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  kg/m^2
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 32.4 (5.5) | 32.5 (5.4) |  |  |  |  | 32.4 (5.5)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 32.7 (5.7) | 32.2 (5.3) | 32.3 (5.5) | 32.6 (5.4) | 32.4 (5.5)
Visual acuity [Mean (Standard Deviation); unit: letters] — Visual acuity is defined as a mean of the acuity scores for both eyes of 74 to 78 letters (the approximate Snellen equivalent of 20/30) Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  letters
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study | 75.9 (10.4) | 75.9 (10.0) |  |  |  |  | 75.9 (10.2)
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies |  |  | 75.6 (10.3) | 75.5 (10.2) | 76.2 (9.7) | 76.2 (10.7) | 75.9 (10.2)
Smoking status [Count of Participants; unit: Participants] — Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  Participants
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study: Never smoked | 581 | 607 |  |  |  |  | 1188
    Glycemic Control Study: Former Smoker | 657 | 623 |  |  |  |  | 1280
    Glycemic Control Study: Current Smoker | 191 | 196 |  |  |  |  | 387
    Glycemic Control Study: Missing | 0 | 1 |  |  |  |  | 1
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies: Never smoked |  |  | 279 | 263 | 313 | 333 | 1188
    Blood Pressure and Lipid Studies: Former Smoker |  |  | 279 | 276 | 373 | 352 | 1280
    Blood Pressure and Lipid Studies: Current Smoker |  |  | 89 | 77 | 119 | 102 | 387
    Blood Pressure and Lipid Studies: Missing |  |  | 0 | 0 | 1 | 0 | 1
Severity of Diabetic Retinopathy [Count of Participants; unit: Participants] — Diabetic retinopathy status was defined according to the eye with the highest level on the ETDRS Final Severity Scale for Persons, as follows: no diabetic retinopathy, a level of less than 20; mild diabetic retinopathy, a level of 20; moderate nonproliferative diabetic retinopathy (NPDR), a level above 20 but less than 53; severe diabetic retinopathy, a level of 53 but less than 60; and proliferative diabetic retinopathy (PDR), a level of 60 or higher. Population: All participants were enrolled in either the intensive or standard glycemia control arms. In addition, participants were included as either part of the blood pressure trial (randomized to intensive or standard) OR the lipid trial (fibrate or fibrate placebo). We completed analysis on participants for whom we had baseline and follow-up data.
  Participants
    Glycemic Control Study: number analyzed (Participants) | 1429 | 1427 | 0 | 0 | 0 | 0 | 2856
    Glycemic Control Study: None | 729 | 721 |  |  |  |  | 1450
    Glycemic Control Study: Mild | 241 | 277 |  |  |  |  | 518
    Glycemic Control Study: Moderate Nonproliferative Diabetic Retinopathy | 443 | 404 |  |  |  |  | 847
    Glycemic Control Study: Severe Nonproliferative Diabetic Retinopathy | 5 | 5 |  |  |  |  | 10
    Glycemic Control Study: Proliferative diabetic retinopathy | 10 | 19 |  |  |  |  | 29
    Glycemic Control Study: Missing | 1 | 1 |  |  |  |  | 2
    Blood Pressure and Lipid Studies: number analyzed (Participants) | 0 | 0 | 647 | 616 | 806 | 787 | 2856
    Blood Pressure and Lipid Studies: None |  |  | 328 | 295 | 429 | 398 | 1450
    Blood Pressure and Lipid Studies: Mild |  |  | 105 | 117 | 141 | 155 | 518
    Blood Pressure and Lipid Studies: Moderate Nonproliferative Diabetic Retinopathy |  |  | 195 | 198 | 230 | 224 | 847
    Blood Pressure and Lipid Studies: Severe Nonproliferative Diabetic Retinopathy |  |  | 3 | 1 | 2 | 4 | 10
    Blood Pressure and Lipid Studies: Proliferative diabetic retinopathy |  |  | 14 | 5 | 4 | 6 | 29
    Blood Pressure and Lipid Studies: Missing |  |  | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression of Diabetic Retinopathy of at Least 3 Stages on the Early Treatment Diabetic Retinopathy Study (ETDRS) Scale, or Development of Proliferative Diabetic Retinopathy Necessitating Photocoagulation Therapy or Vitrectomy
Description: Diabetic retinopathy status was defined according to the eye with the highest level on the ETDRS Final Severity Scale for Persons, as follows: no diabetic retinopathy, a level of less than 20; mild diabetic retinopathy, a level of 20; moderate nonproliferative diabetic retinopathy (NPDR), a level above 20 but less than 53; severe diabetic retinopathy, a level of 53 but less than 60; and proliferative diabetic retinopathy (PDR), a level of 60 or higher.
Time Frame: Measured at Year 4
Population: The ACCORD Eye study recruited 3472 eligible participants. Of these, 2856 participants had both baseline and year 4 follow-up data available for analyses.
Measure: Number; unit: participants
Groups:
- Intensive Glycemia Control: Strategy of intensive glycemia treatment to HbA1c less than 6%
- Standard Glycemia Control: Strategy of multiple drugs to treat HbA1c to 7.0% - 7.9%
- Intensive Blood Pressure Control: A strategy of BP treatment for SBP less than 120 mmHg
- Standard Blood Pressure Control: Strategy of BP treatment for SBP less than 140 mmHg
- Fenofibrate + Simvastatin Therapy: Blinded fenofibrate + simvastatin 20-40 mg/d
- Placebo + Simvastatin Therapy: Blinded placebo + simvastatin 20-40 mg/d
Arm/Group | Intensive Glycemia Control | Standard Glycemia Control | Intensive Blood Pressure Control | Standard Blood Pressure Control | Fenofibrate + Simvastatin Therapy | Placebo + Simvastatin Therapy
Number analyzed (Participants) | 1429 | 1427 | 647 | 616 | 806 | 787
participants | 104 | 149 | 67 | 54 | 52 | 80
Statistical Analysis 1: Comparison: Intensive Glycemia Control vs Standard Glycemia Control; Our recruitment goal for the ACCORD Eye study was set in order to achieve a statistical power of 88% to detect a 15% relative reduction with intensive glycemic control as compared with standard glycemic control; Test type: Superiority or Other; p = 0.003, Regression, Logistic; Comparisons made using likelihood-ratio tests from logistic-regression models with adjustment for same study-design factors used in ACCORD analysis; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.51 to 0.87]
Statistical Analysis 2: Comparison: Intensive Blood Pressure Control vs Standard Blood Pressure Control; Our recruitment goal for the ACCORD Eye study was set in order to achieve a statistical power of 80% to detect a 20% relative reduction with intensive blood pressure control as compared with standard blood pressure control; Test type: Superiority or Other; p = 0.29, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.84 to 1.79]
Statistical Analysis 3: Comparison: Fenofibrate + Simvastatin Therapy vs Placebo + Simvastatin Therapy; Our recruitment goal for the ACCORD Eye study was set in order to achieve a statistical power of 91% to detect a 20% relative reduction with lipid control with a statin and fenofibrate as compared with lipid control with a statin alone; Test type: Superiority or Other; p = 0.006, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.42 to 0.87]

2. Secondary Outcome: Loss of Visual Acuity
Time Frame: Measured at Year 4
Population: Subset of Participants from the entire ACCORD cohort (NCT00000620) who provided information about loss in visual acuity.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Glycemia Control | Standard Glycemia Control | Intensive Blood Pressure Control | Standard Blood Pressure Control | Fenofibrate + Simvastatin Therapy | Placebo + Simvastatin Therapy
Number analyzed (Participants) | 3466 | 3511 | 1629 | 1617 | 1883 | 1848
Participants | 744 | 752 | 367 | 382 | 354 | 393
Statistical Analysis 1: Comparison: Intensive Glycemia Control vs Standard Glycemia Control; Test type: Superiority or Other; p = 0.96, Regression, Cox; Hazard Ratio (HR) = 0.997, 95% CI 2-sided [0.901 to 1.104]
Statistical Analysis 2: Comparison: Intensive Blood Pressure Control vs Standard Blood Pressure Control; Test type: Superiority or Other; p = 0.50, Regression, Cox; Hazard Ratio (HR) = 0.952, 95% CI 2-sided [0.825 to 1.099]
Statistical Analysis 3: Comparison: Fenofibrate + Simvastatin Therapy vs Placebo + Simvastatin Therapy; Test type: Superiority or Other; p = 0.08, Regression, Cox; Hazard Ratio (HR) = 0.880, 95% CI 2-sided [0.762 to 1.016]

3. Secondary Outcome: Cataract Extraction
Time Frame: Measured at Year 4
Population: Subset of Participants from the entire ACCORD cohort (NCT00000620) who provided information regarding whether or not they had a cataract extraction.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Glycemia Control | Standard Glycemia Control | Intensive Blood Pressure Control | Standard Blood Pressure Control | Fenofibrate + Simvastatin Therapy | Placebo + Simvastatin Therapy
Number analyzed (Participants) | 4361 | 4405 | 2053 | 2039 | 2333 | 2341
Participants | 547 | 623 | 266 | 300 | 305 | 299
Statistical Analysis 1: Comparison: Intensive Glycemia Control vs Standard Glycemia Control; Test type: Superiority or Other; p = 0.0355, Regression, Cox; Hazard Ratio (HR) = 0.884, 95% CI 2-sided [0.788 to 0.992]
Statistical Analysis 2: Comparison: Intensive Blood Pressure Control vs Standard Blood Pressure Control; Test type: Superiority or Other; p = 0.17, Regression, Cox; Hazard Ratio (HR) = 0.891, 95% CI 2-sided [0.755 to 1.051]
Statistical Analysis 3: Comparison: Fenofibrate + Simvastatin Therapy vs Placebo + Simvastatin Therapy; Test type: Superiority or Other; p = 0.86, Regression, Cox; Hazard Ratio (HR) = 1.015, 95% CI 2-sided [0.865 to 1.190]

4. Secondary Outcome: Development or Progression of Macular Edema
Time Frame: Measured at Year 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Glycemia Control | Standard Glycemia Control | Intensive Blood Pressure Control | Standard Blood Pressure Control | Fenofibrate + Simvastatin Therapy | Placebo + Simvastatin Therapy
Number analyzed (Participants) | 1413 | 1399 | 633 | 609 | 791 | 779
Participants | 44 | 40 | 18 | 20 | 24 | 22
Statistical Analysis 1: Comparison: Intensive Glycemia Control vs Standard Glycemia Control; Test type: Superiority or Other; p = 0.069, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.71 to 1.69]
Statistical Analysis 2: Comparison: Intensive Blood Pressure Control vs Standard Blood Pressure Control; Test type: Superiority or Other; p = 0.63, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.44 to 1.63]
Statistical Analysis 3: Comparison: Fenofibrate + Simvastatin Therapy vs Placebo + Simvastatin Therapy; Test type: Superiority or Other; p = 0.78, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.60 to 1.96]

ADVERSE EVENTS:
Time Frame: Entire duration of the study
Description: Adverse events were collected as part of the ACCORD main trial (NCT00000620). No adverse events were collected as part of the ACCORD-Eye Study.
Arm/Group | Intensive Glycemia Control | Standard Glycemia Control | Intensive BP Control | Standard BP Control | Fibrate | Fibrate Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The glycemia trial was stopped early, potentially underestimating the reported effect of glycemia treatment on diabetic retinopathy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No